CLINICAL TRIAL: NCT05195073
Title: Three Dimensional Versus Two-dimensional Laparoscopic Salpingectomy in Patients With Hydrosalpinx Undergoing IVF-ET. A Randomized Controlled Trial
Brief Title: Three Dimensional Versus Two Dimensional Laparoscopic Salpingectomy in Patients With Hydrosalpinx Undergoing IVF-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abdalla, lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D Laparoscopic salpingectomy
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Hydrosalpinx
Keywords: Hydrosalpinx; Infertility; In vitro fertilization; Laparoscopy
MeSH Terms: conditions — Infertility | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 D laparoscopy group (Active Comparator): salpingectomy will be performed by using Storz image 1 S 3D laparoscopy system (Karl Storz, Tuttlingen, Germany) which is comprised of a 10 mm scope with 2 full HD sensors at the tip of the scope and a 3 D control unit plus a 3 D display
  Interventions: Biological: Laparoscopy
- 2 D laparoscopy group (Active Comparator): salpingectomy will be performed by using a conventional 2 D laparoscopy system.
  Interventions: Biological: Laparoscopy

INTERVENTIONS:
Biological: Laparoscopy — 3 D laparoscopy

SUMMARY:
A three-dimensional laparoscopic vision system (3-D LVS) has gained acceptance and is being utilized in daily practice despite debates about its success.

DETAILED DESCRIPTION:
A three-dimensional laparoscopic vision system (3-D LVS) has gained acceptance and is being utilized in daily practice despite debates about its success. in our study we will compare operative data and early postoperative outcomes of laparoscopic salpingectomy operations conducted using standard 2-D and 3-D laparoscopic vision systems

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral hydrosalpinx diagnosed with hysterosalpingography or laparoscopy

Exclusion Criteria:

* Bilateral hydrosalpinx,
* co-existent adnexal pathology,
* body mass index (BMI) more than 40,
* extensive pelvic adhesions,
* coagulation defects or concurrent anticoagulant therapy,
* compromised cardiopulmonary status,
* and contraindications for general anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The time required to excise the hydrosalpinx | 6 months
  The time required to excise the hydrosalpinx

SECONDARY OUTCOMES:
The degree of difficulty experienced by the surgeon | 6 months
  The degree of difficulty experienced by the surgeon during excision of the hydrosalpinx [ evaluated using a visual analog scale ranging from 0 (least difficult) to 10 (most difficult)].
The total operative time. | 6 months
  The total operative time.
The amount of Intraoperative blood loss. | 6 months
  The amount of Intraoperative blood loss.
Rate of intraoperative and postoperative complications. | 6 months
  Rate of intraoperative and postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Abdalla, Principal Investigator — Kasralainy teaching hospital
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fouda UM, Sayed AM. Effect of ultrasound-guided aspiration of hydrosalpingeal fluid during oocyte retrieval on the outcomes of in vitro fertilisation-embryo transfer: a randomised controlled trial (NCT01040351). Gynecol Endocrinol. 2011 Aug;27(8):562-7. doi: 10.3109/09513590.2010.507290. Epub 2010 Jul 30. PMID 20672903
- [Background] Strandell A, Lindhard A, Waldenstrom U, Thorburn J, Janson PO, Hamberger L. Hydrosalpinx and IVF outcome: a prospective, randomized multicentre trial in Scandinavia on salpingectomy prior to IVF. Hum Reprod. 1999 Nov;14(11):2762-9. doi: 10.1093/humrep/14.11.2762. PMID 10548619
- [Background] Fouda UM, Sayed AM, Abdelmoty HI, Elsetohy KA. Ultrasound guided aspiration of hydrosalpinx fluid versus salpingectomy in the management of patients with ultrasound visible hydrosalpinx undergoing IVF-ET: a randomized controlled trial. BMC Womens Health. 2015;15:21. doi: 10.1186/s12905-015-0177-2. Epub 2015 Feb 27. PMID 25783650
- [Background] Johnson N, van Voorst S, Sowter MC, Strandell A, Mol BW. Surgical treatment for tubal disease in women due to undergo in vitro fertilisation. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD002125. doi: 10.1002/14651858.CD002125.pub3. PMID 20091531
- [Background] Fouda UM, Elsetohy KA, Elshaer HS. Barbed Versus Conventional Suture: A Randomized Trial for Suturing the Endometrioma Bed After Laparoscopic Excision of Ovarian Endometrioma. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):962-8. doi: 10.1016/j.jmig.2016.06.008. Epub 2016 Jun 18. PMID 27329547